CLINICAL TRIAL: NCT05051124
Title: PT4A (Peers and Technology for Adherence, Access, Accountability, and Analytics) - A Qualitative Study
Brief Title: Peers and Technology for Adherence, Access, Accountability, and Analytics
Acronym: PT4A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-01579; 1R56HL150036 (NIH)
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Medication Adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Enrolled in the AMPATH CDM Program (Experimental)
  Interventions: Behavioral: Peer Delivery of Medications; Behavioral: Health Information Technology (HIT) Platform

INTERVENTIONS:
Behavioral: Peer Delivery of Medications — The study team will adopt a novel approach of extending beyond the use of peer support in the clinical setting and implement door-to-door peer delivery of medications within patients' communities
Behavioral: Health Information Technology (HIT) Platform — To support peer delivery, the study team will use a HIT platform that performs 4 core functions: 1) tailored counseling strategies through decision support; 2) teleconsultation support for clinician-peer-patient interactions; 3) tracking medication refills to enhance accountability of the peer delivery process; and 4) analytics to improve medication supply chain by generating patient-level drug consumption data. This is an innovative use of HIT to accomplish these functions to support medication adherence.

SUMMARY:
The overall objective of this project is to utilize the PRECEDE-PROCEED framework to conduct transdisciplinary, translational implementation research focused on improving medication adherence for hypertension control. The central hypothesis is that peer delivery of medications integrated with HIT (PT4A) will be effective in improving hypertension medication adherence, contributing to improved blood pressure among patients with uncontrolled hypertension in western Kenya. This study record will focus on Sub-Aim 2.2: a pilot of the intervention and a survey questionnaire with patients, peers, and clinical staff to evaluate feasibility. The investigators will evaluate impact on systolic blood pressure, medication adherence, and fidelity of implementation. The investigators will also create a retrospective comparator (control) group of CDM patients, through querying AMRS, matched by sex, age, location and initial blood pressure level. The investigators will then use their recorded blood pressure over a comparable period of up to 1 year and to allow for comparison to the blood pressure changes observed in the patients enrolled in the PT4A program to help understand the magnitude and variance of the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Enrolled in the AMPATH CDM PRogram
* Have uncontrolled hypertension (defined as systolic blood pressures ≥ 140 or diastolic blood pressure ≥ 90)

Exclusion Criteria:

* Acute illness requiring immediate medical attention
* Terminal illness
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Vedanthan, MD, MPH, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose will have access to the data upon reasonable request. Requests should be directed to rajesh.vedanthan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Enrolled in the AMPATH CDM Program
Started | 101
Completed | 95
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Residential relocation | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Enrolled in the AMPATH CDM Program
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 95
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 95

OUTCOME MEASURES:

1. Primary Outcome: Absolute Mean Change in Systolic Blood Pressure (SBP)
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Patients Enrolled in the AMPATH CDM Program
Number analyzed (Participants) | 95
millimeters of mercury (mmHg) | 11.5 (23.9)

2. Primary Outcome: Pill Count Adherence Ratio
Description: Proportion of prescribed doses taken over a 1-month time period.
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: Proportion of prescribed doses
Arm/Group | Patients Enrolled in the AMPATH CDM Program
Number analyzed (Participants) | 95
Proportion of prescribed doses | 0.99 (0.08)

3. Primary Outcome: Number of Confirmed Medication Deliveries
Description: Confirmed medication delivery will be documented by patient e-signature.
Time Frame: Month 12
Measure: Number; unit: Deliveries
Arm/Group | Patients Enrolled in the AMPATH CDM Program
Number analyzed (Participants) | 101
Deliveries | 992

4. Primary Outcome: Number of Peer Completions of HIT Form
Time Frame: Month 12
Measure: Number; unit: Completed forms
Arm/Group | Patients Enrolled in the AMPATH CDM Program
Number analyzed (Participants) | 101
Completed forms | 999

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Patients Enrolled in the AMPATH CDM Program
All-Cause Mortality (participants affected / at risk) | 1/101
Serious Adverse Events (participants affected / at risk) | 1/101
Other Adverse Events (participants affected / at risk) | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Enrolled in the AMPATH CDM Program (N=101)
Death (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT05051124/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT05051124/ICF_000.pdf